CLINICAL TRIAL: NCT06306105
Title: Assessment of Anti-aging Efficacy of Marine Collagen Peptides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23-118-B
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Skin Condition; Hair Fragility; Nails, Ingrown
Keywords: fish collagen
MeSH Terms: conditions — Skin Diseases; Nails, Ingrown

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: placebo drink
- Marine Collagen Peptides drinks (Experimental)
  Interventions: Dietary Supplement: Marine Collagen Peptides

INTERVENTIONS:
Dietary Supplement: Marine Collagen Peptides — consume 1 bottle per day
  Other Names: Coral club Promarine Collagen Tripeptides
  Arms: Marine Collagen Peptides drinks
Dietary Supplement: placebo drink — consume 1 bottle per day
  Arms: placebo drink

SUMMARY:
To assess the anti-aging efficacy of Marine Collagen Peptides on skin, hair and finger nails for human

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged above 18 years old

Exclusion Criteria:

* Subjects who are not volunteers
* Subjects who have been diagnosed with dermatitis, cirrhosis, and chronic kidney failure
* Subjects who have known cosmetic, drug or food allergies.
* Patients are taking medicine for chronic diseases
* Subjects receiving treatments for scalp, hair transplant, and other scalp medical care in past 12 weeks.
* Subjects getting a manicure and perm in past 12 weeks.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Subjects receiving facial laser therapy, chemical peeling or UV overexposure (> 3 hr/week) in the past 12 weeks.
* Students who are currently taking courses taught by the principal investigator of this trial.
* Subjects are not willing to reveal the results of pictures after taking the product
* Vegetarian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
The change of skin hydation | Change from Baseline skin skin hydation at 12 weeks
  Corneometer® CM825 (CK, Germany) was utilized to measure skin surface hydation. Units: arbitrary Corneometer® units 0-120.
The change of skin wrinkles | Change from Baseline skin wrinkles at 12 weeks
  VISIA Complexion Analysis was utilized to measure skin wrinkles. Units: the amount of detectable wrinkles
The change of skin elasticity | Change from Baseline skin elasticity at 12 weeks
  Cutometer® MPA580 was utilized to measure skin elasticity. Units: visco-elasticity in %.
The change of skin collagen density | Change from Baseline skin collagen density at 12 weeks
  DermaLab® Series SkinLab Combo was utilized to measure skin collagen density. Units: arbitrary units
The change of hair diameters | Change from Baseline hair diameters at 12 weeks
  Mitutoyo C/N293-100 was utilized to measure hair diameters. Units: millimeter
The change of hair loss amount | Change from Baseline hair loss amount at 12 weeks
  Collect and measure the weight of loss hair. Units: gram
The change of hair roots diameters | Change from Baseline hair roots diameters at 12 weeks
  Mitutoyo C/N293-100 was utilized to measure hair roots diameters. Units: millimeter
The change of hair density | Change from Baseline hair density at 12 weeks
  Soft Plus was utilized to picture and observe hair density.
The change of hair follicle strength | Change from Baseline hair follicle strength at 12 weeks
  Pull up the hair of the frontal bone, temporal bone and occipital bone (approximately 60 hairs/area) to assess the number of hair loss in each area. Units: the number of loss hair
The change of thumbs nail color | Change from Baseline thumbs nail color at 12 weeks
  Chroma Meter MM500 was utilized to measure thumbs nail color. Units: L* index
The change of nails appearence | Change from Baseline nails appearence at 12 weeks
  Picture taken was utilized to record and observe nails appearence.
The change of nails growth | Change from Baseline marking position at 12 weeks
  Marking the position of middle fingers lunula was utilized to record and observe nails growth. Units: milimeter
The degree of nails fragility | Change from Baseline nails fragility at 12 weeks
  Iron ruler was utilized to evaluate nails fragility. Picture taken was utilized to record and observe the change of nails fragility.

SECONDARY OUTCOMES:
The change of self-assessment skin, hair, and nails condition | Change from Baseline skin, hair, and nails condition at 12 weeks
  A self-assessment questionnaire was collected and evaluate skin, hair, and nails condition

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Ph.D., Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy & Science, Pingtung City, Taiwan